CLINICAL TRIAL: NCT06433934
Title: Comparison of the Oxymask and Oxy2mask on Supplemental Oxygen Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Patti DeJuilio, Director Respiratory Care and Diagnostic Services, Northwestern Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oxymask
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Each patient will receive mask #1, then receive mask #2. The flowrate to maintain same desired oxygen saturations will be documented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Oxy2mask (Experimental): Change oxymask to oxy2mask
  Interventions: Device: Oxy2mask

INTERVENTIONS:
Device: Oxy2mask — Open design oxygen mask

SUMMARY:
The purpose of this study is to determine if the performance of a newly released oxygen mask is the same, better, or worse than previous mask version. We will measure the flow rate necessary to maintain the same oxygen saturation in adult patients using each mask.

DETAILED DESCRIPTION:
Southmedic, Inc. has received approval to distribute a newly designed oxygen mask. The current design has been studied and the FiO2 delivered reported to be inconsistent. The purpose of this study is to determine if the performance is the same, better, or worse than current mask. We can evaluate performance by determining Liter flow required to maintain oxygen saturations that are within limits described in NM CDH oxygen protocol. We will measure the flow rate necessary to maintain the same saturation in adult patients using both the OxyMask and Oxy2Mask. The Oxymask has a flow device inside the mask that has been revised since implementation. The mask itself is otherwise unchanged. We intend to determine if the same amount of flow results in the same outcome.

This study will include adult patients that require supplemental oxygen and we do not believe the patients will report a difference between each mask. The only variance in care is mask version used, the oxygen protocol will remain the same.

ELIGIBILITY:
Inclusion Criteria:

* Participants have oxygen device and are being titrated per NM CDH oxygen protocol (maintained between 90%-96%; or 88% - 92% if CO2 retainer)
* Participants to have period of stability; 2 hours at same liter flow on open design mask, 5-15 lpm 02.
* All adult patients (> 18 years old) in med surge units (bed tower)
* Post-op patients requiring oxygen on Post-op Day 2.
* Patients currently on >5 LPM via nasal cannula, clinician can recommend the change to OxyMask. If remains on >5 LPM via OxyMask, patient can be included.
* Oxygen protocol will be followed per standards of care.

Exclusion Criteria:

* Patients receiving home oxygen therapy who do not require additional oxygen during hospital stay.
* Patients with a history of Bleomycin therapy.
* Patients with a history of Paraquat poisoning
* Patients that are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Required Flowrate | 4 hours
  Flow (LPM) required to maintain target oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Megan Carney, Study Director — Northwestern Medicine IRB
Locations (1):
- Central DuPage Hospital, Winfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No